CLINICAL TRIAL: NCT03104478
Title: Real Time Molecular Characterization of Diffuse Large B Cell Lymphoma (DLBCL)
Acronym: RT3
Status: Completed | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: RT3
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL; Real time molecular characterization
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected at time of enrollment in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biological samples collection — In addition to collection and characterization of tumor biopsy samples done for diagnosis (standard care), collection of blood samples at study entry for further biological analyses.

SUMMARY:
The trial will enroll 194 previously untreated DLBCL patients over 20 months, with the objective to send to the local investigator an extensive molecular tumor characterization by D38 in at least 80% of enrolled patients.

The feasibility and efficiency will be demonstrated by deploying and operating a nation-wide network of dedicated multidisciplinary platforms.

ELIGIBILITY:
Inclusion Criteria:

* DLBCL patients that will be eligible in front-line treatment for a combination of anthracycline-based chemotherapy plus anti-CD20 monoclonal antibody,Rituximab: R-CHOP 14, R-CHOP 21, R mini-CHOP, R-ACVBP, R-COPADEM. Patients treated with R-CHOP associated with an experimental drug ((polatuzumab, tazemetostat, venetoclax, entospletinib, lenalidomide, ibrutinib, anti PD1/anti PDL1 ….)
* A short corticotherapy (prednisone, maximum 7 days) given during pre-phase therapy is allowed.
* Eligible histological subtypes: in particular DLBCL NOS, PMBL, high grade B-cell lymphoma (HGBCL) withMYC and BCL2 and/or BCL6 rearrangements, HGBCL NOSFL grade 3B and untreated transformed low grade NHL.
* ≥ 18 years old, IPI = 0-5
* With available tumor Biopsy (FFPE) that can be sent to RT3 platform at the time of inclusion (or the say after inclusion at the latest).
* Patient that underwent needle core biopsy samples are not excluded if sufficient material is available for molecular and histopathological explorations

Exclusion Criteria:

* No available FFPE biopsy material or insufficient quality/quantity tumor samples according to prerequisite
* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient ≥ 18 years old with prior untreated DLBCL
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
Real time report of molecular characterization | 38 days (i.e. 38 days after starting inductive chemotherapy regimen
  To timely report the molecular characterization (pathogenic, diagnostic, prognostic, theranostic markers) of previously untreated DLBCL patients prior to day 38(i.e. 38 days after starting inductive chemotherapy regimen, in at least 80% of enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jardin, Pr, Principal Investigator — Lymphoma Study Association; Christiane Copie, Pr, Principal Investigator — Lymphoma Study Association
Locations (15):
- France (15):
  - CHU Caen, Caen
  - Hopital Henri Mondor, Créteil
  - CHU Le Bocage, Dijon
  - CH Départemental, La Roche-sur-Yon
  - CHU Claude Hurriez, Lille
  - CHU Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Centre Francois Magendie, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de la Miletrie, Poitiers
  - Ch Annecy Genevois, Pringy
  - Centre Henri Becquerel, Rouen
  - IUCT Oncopôle - CHU de Toulouse, Toulouse
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No